CLINICAL TRIAL: NCT02949440
Title: A Prospective Randomized Controlled Clinical Study of Laparoscopic Right Hemicolectomy Using the Caudal-to-cranial Approach
Brief Title: A Study of Laparoscopic Right Hemicolectomy Using the Caudal-to-cranial Approach
Acronym: LRHCTC-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liao-nan Zou,Prof, professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LRHCTC-1
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Ascending Colon Cancer; Ileocaecal Valve Carcinoma; Cancer Flexure Hepatic; Adenocarcinoma of Hepatic Flexure (Diagnosis)
Keywords: Laparoscopic right Hemicolectomy; Caudal-to-cranial Approach
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the caudal-to-cranial approach (Experimental): Cutting the peritoneum along the line between the right mesocolon and retroperitoneum, enter the Toldt's space to dissect the posterior of Superior mesenteric vein（SMV）and Superior mesenteric artery（SMA）and their branches, and then finished the D3 dissection from caudal to cranial on both sides of the mesentery along the Superior mesenteric vein（SMV）. In the end, cut the lateral ligament to mobilize the posterior space of ascending colon. This approach is called caudal-to-cranial approach.
  Interventions: Procedure: the caudal-to-cranial approach
- the medial-to-lateral approach (Active Comparator): First, the pedicle of ileocolic vessels is identified and the mesocolon is dissected between the pedicle and the periphery of the Superior mesenteric vein（SMV）to expose the second portion of the duodenum. The ileocolic vessels are then cut at their roots. The ascending mesocolon is separated from the retroperitoneal tissues, duodenum, and pancreatic head up to the hepatocolic ligament cranially. The important detail in this procedure is the wide separation between the pancreatic head and the transverse mesocolon.This approach is the medial-to-lateral(MtL) approach
  Interventions: Procedure: the medial-to-lateral approach

INTERVENTIONS:
Procedure: the caudal-to-cranial approach — Cutting the peritoneum along the line between the right mesocolon and retroperitoneum, enter the Toldt's space to dissect the posterior of Superior mesenteric vein and Superior mesenteric artery and their branches, and then finished the D3 dissection from caudal to cranial on both sides of the mesentery along the Superior mesenteric vein. In the end, cut the lateral ligament to mobilize the posterior space of ascending colon. This approach is called the caudal-to-cranial approach.
  Arms: the caudal-to-cranial approach
Procedure: the medial-to-lateral approach — First, the pedicle of ileocolic vessels is identified and the mesocolon is dissected between the pedicle and the periphery of the Superior mesenteric vein to expose the second portion of the duodenum. The ileocolic vessels are then cut at their roots. The ascending mesocolon is separated from the retroperitoneal tissues, duodenum, and pancreatic head up to the hepatocolic ligament cranially. The important detail in this procedure is the wide separation between the pancreatic head and the transverse mesocolon.This approach is the medial-to-lateral(MtL) approach
  Arms: the medial-to-lateral approach

SUMMARY:
To investigate the clinical application value of laparoscopic radical right hemicolectomy using the caudal-to-cranial approach versus the medial-to-lateral approach by prospective randomized controlled clinical study.

DETAILED DESCRIPTION:
To compare the caudal-to-cranial approach with the medial-to-lateral approach in laparoscopic right hemicolectomy for the advance right colon cancer.

A prospective randomized controlled trial will be performed in the GI department,the Guangdong provincial hospital of Chinese Medicine from October 2016 to October 2024.The sample size，150 cases with advanced right colon cancer, will be needed after calculated by the statistics .The 150 cases will be randomly divided into two groups: laparoscopic radical right hemicolectomy using the caudal-to-cranial(CtC) approach(GroupCtC) and laparoscopic radical right hemicolectomy using the medial-to-lateral(MtL) approach (GroupMtL). Primary outcomes are the operative time，The secondary outcomes are the total blood loss,the number of lymph nodes dissected,the average time of ground activities,the time to first flatus,the hospital stay,the intra-operative complication and the post-operative complication，and others' outcomes are the Disease-free survival rate(DFS) at 3 years and 5 years,the Overall survival rate（OS）at 3 years and 5 years.The data in two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. The age limits is 18-80 years old;
2. The clinical staging was II,III carcinoma of right colon，located in right-sided colon;
3. The preoperative imaging confirmed that the tumor did not involve adjacent organs;
4. American Society of anesthesiologists (ASA) score less than or equal to Level III;
5. Criteria of performance status karnofsky is greater than or equal to 60.

Exclusion Criteria:

1. The patients' age limits is Less than 18 years old, or more than 80 years old
2. The preoperative imaging confirmed that the tumor involve adjacent organs;
3. The tumor have been finding distant metastases;
4. American Society of anesthesiologists (ASA) score more than 3;
5. Criteria of performance status karnofsky is lower than 60;
6. It is the carcinoma of right colon with multiple colonic polyps Disease;
7. there is a laparoscopic surgery contraindications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the operation time | up to 36 months

SECONDARY OUTCOMES:
the total blood loss | up to 36 months
the number of lymph nodes dissected | up to 36 months
the average time of ground activities | up to 36 months
the time to first flatus | up to 36 months
the intra-operative complication and the post-operative complication | up to 36 months

OTHER OUTCOMES:
the 3-year and 5-year Disease-free survival（DFS） | up to 3 years and 5 years
3-year and 5-year Overall survival（OS） | up to 3 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Liao-nan Zou, professor, Principal Investigator — GI surgery,Guangdong Province Hospital of Chinese Medicine; Jin Wan, PhD, Study Director — GI surgery,Guangdong Province Hospital of Chinese Medicine
Locations (1):
- GI surgery,Guangdong Province Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Zou L, Xiong W, Li H, He Y, Diao D, Zheng Y, Luo L, Tan P, Wang W, Wan J. [Efficacy analysis of laparoscopic radical right hemicolectomy using caudal-to-cranial approach]. Zhonghua Wei Chang Wai Ke Za Zhi. 2015 Nov;18(11):1124-7. Chinese. PMID 26616807
- [Result] Zou L, Xiong W, Mo D, He Y, Li H, Tan P, Wang W, Wan J. Laparoscopic Radical Extended Right Hemicolectomy Using a Caudal-to-Cranial Approach. Ann Surg Oncol. 2016 Aug;23(8):2562-3. doi: 10.1245/s10434-016-5215-2. Epub 2016 Apr 12. PMID 27072997
- [Result] Li H, He Y, Lin Z, Xiong W, Diao D, Wang W, Wan J, Zou L. Laparoscopic caudal-to-cranial approach for radical lymph node dissection in right hemicolectomy. Langenbecks Arch Surg. 2016 Aug;401(5):741-6. doi: 10.1007/s00423-016-1465-5. Epub 2016 Jun 18. PMID 27318491